CLINICAL TRIAL: NCT00947531
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Safety and Efficacy of 20 ml Cerebrolysin in Patients With Vascular Dementia
Brief Title: A Clinical Trial to Evaluate the Safety and Efficacy of 20 ml Cerebrolysin in Patients With Vascular Dementia
Acronym: VascDem
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ever Neuro Pharma GmbH (Industry)
Collaborators: acromion GmbH (Industry); Geny Research Corp. (Unknown)
Responsible Party: Philipp Novak, PhD, EBEWE Neuro Pharma
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EBE-RU-051201
Record Dates: First submitted 2009-04-20; First posted 2009-07-28 (Estimated); Results first posted 2009-07-28 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Vascular Dementia
MeSH Terms: conditions — Dementia, Vascular | interventions — cerebrolysin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cerebrolysin (Experimental)
  Interventions: Drug: Cerebrolysin
- 0.9% Saline Solution (Placebo Comparator)
  Interventions: Drug: 0.9% Saline Solution

INTERVENTIONS:
Drug: Cerebrolysin
  Arms: Cerebrolysin
Drug: 0.9% Saline Solution
  Arms: 0.9% Saline Solution

SUMMARY:
This clinical trial was performed to assess the clinical efficacy and safety of two 4 week treatment courses of daily intravenous administration of Cerebrolysin (20mL [milliliter] IV [intravenous] per day). The study was performed as prospective, randomised, double-blind, placebo-controlled, parallel group, multicentre study with 2 study groups.

Group 1: 20 mL Cerebrolysin and 100 mg (milligram) acetylsalicylic acid Group 2: Placebo (0.9% NaCl [sodium chloride]) and 100 mg acetylsalicylic acid The study drug was given once daily by intravenous infusion (20ml in 250ml saline solution) for 4 weeks on five consecutive days per week. This treatment regimen was repeated after a two-month treatment-free interval. Acetylsalicylic acid was given orally, once daily throughout the study duration of 24 weeks.

Altogether five clinical evaluation visits at Baseline (day 0) and at week 4, 12, 16, and 24 were necessary.

ELIGIBILITY:
Inclusion Criteria:

* Men or post-menopausal women between 50 and 85 years
* Clinical diagnosis of vascular dementia according to NINDS-AIREN criteria
* CT or MRI results compatible with clinical diagnosis
* MMSE score between 10 and 24, both inclusive
* Modified Hachinski Ischemic Score >4
* Hamilton Depression Scale score of less than or equal to 15
* Adequate visual and auditory acuity to allow neuropsychological testing
* Informed consent given by the patient and/or the next-of-kin

Exclusion Criteria:

* Gastric ulcer associated with intolerance of acetylsalicylic acid treatment
* Severe psychotic features, schizophrenia, depression, agitation or behavioral problems within the last three months that could lead to difficulty complying with the protocol
* Any severe systemic illness or unstable medical condition that could lead to difficulty complying with the protocol or significantly limits life span.
* Patients who in the investigator's opinion, would not comply with study procedures
* Any significant neurological disease other than vascular dementia, such as Parkinson's disease, epilepsy, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, or multiple sclerosis
* History of alcohol or substance abuse or dependence within the past two years
* Patients with a history of systemic cancer within the past two years
* Severe congestive heart failure or malignant, uncontrollable hypertension
* Participation in a clinical trial with an investigational drug in the past four weeks

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2006-10; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Novak, PhD, Study Director — EBEWE Neuro Pharma
Locations (21):
- Russia (21):
  - Chita State Medical Academy/Regional Psychiatric Hospital No. 2, Chita
  - Chita State Medical Academy/Veterans Hospital, Chita
  - Irkutsk State Institute of Postgraduate Education/Regional Clinical Hospital, Irkutsk
  - Kazan State Medical University/Municipal Clinical Hospital No. 6, Kazan'
  - Kazan State Medical University/Republican Clinical Hospital, Kazan'
  - Kursk Medical University/Kursk Regional Clinical Hospital, Kursk
  - I. M. Sechenov Moscow Medical Academy, Moscow
  - Mental Health Research Center of RAMS/Psychiatric Clinical Hospital No. 15, Moscow
  - Mental Health Research Center of RAMS, Moscow
  - Russian Medical Academy of Postgraduate Education/S. P. Botkin Municipal Clinical Hospital, Moscow
  - Russian State Medical University/N. I. Pirogov Municipal Clinical Hospital No. 1, Moscow
  - Scientific Research Institute of Neurology of RAMS, Moscow
  - Municipal Clinical Hospital No. 5, Nizhny Novgorod
  - N. A. Semashko Nizhniy Novgorod Regional Clinical Hospital, Nizhny Novgorod
  - Central Municipal Hospital, Reutov
  - I. P. Pavlov St. Petersburg State Medical University, Saint Petersburg
  - S. M. Kirkov Medical Military Academy of the Ministry of Defense of RF, Saint Petersburg
  - V. M. Bekhterev St. Petersburg Scientific Research Psychoneurological Institute, Saint Petersburg
  - Saratov Regional Psychiatric Hospital of Snt. Sofia, Saratov
  - Bashkirian State Medical University/Emergency Medical Care Hospital, Ufa
  - Yaroslavl State Medical Academy/Yaroslavl Clinical Hospital No. 8, Yaroslavl

REFERENCES:
- [Result] Guekht AB, Moessler H, Novak PH, Gusev EI; Cerebrolysin Investigators. Cerebrolysin in vascular dementia: improvement of clinical outcome in a randomized, double-blind, placebo-controlled multicenter trial. J Stroke Cerebrovasc Dis. 2011 Jul-Aug;20(4):310-8. doi: 10.1016/j.jstrokecerebrovasdis.2010.01.012. Epub 2010 Jul 24. PMID 20656516

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of recruitment period: 24-Oct-2006 - 02-Feb-2007 Type of location: Hospitals, Medical Universities, Medical Military Academy, Research Institutes
Pre-assignment Details: Patients were excluded from the trial before assignment to a group when not all inclusion criteria were met or when exclusion criteria were applicable.
Period: Overall Study
Arm/Group | Cerebrolysin | 0.9% Saline Solution
Started | 121 | 121
Completed | 107 | 110
Not Completed | 14 | 11
Not completed — Withdrawal by Subject | 10 | 7
Not completed — Administrative Reason | 0 | 1
Not completed — Adverse Event | 2 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cerebrolysin | 0.9% Saline Solution | Total
Number analyzed (Participants) | 121 | 121 | 242
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 39 | 77
  >=65 years | 83 | 82 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (8.0) | 67.6 (8.0) | 67.3 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 72 | 154
  Male | 39 | 49 | 88
Region of Enrollment [Number; unit: participants]
  Russian Federation | 121 | 121 | 242

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in ADAS-cog+ (Alzheimer's Disease Assesment Scale - Cognitive Subpart) at Week 24
Description: The ADAS-COG+ is a psychometric instrument used to evaluate memory, attention, reasoning, language, orientation and praxis. The score ranges from 0 to 85 with 85 being the worst score. A negative change indicates cognitive improvement.
Time Frame: baseline and week 24
Population: The primary and confirmatory analysis is based on the ITT analysis set. The LOCF method is applied to account for missing data. The ITT analysis set consists of all randomized patients, who received at least one dose of study medication and had a baseline and at least one post-baseline assessment for both primary efficacy measures.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Cerebrolysin | 0.9% Saline Solution
Number analyzed (Participants) | 117 | 115
points on a scale | -10.60 (7.77) | -4.49 (8.13)
Statistical Analysis 1: Comparison: Cerebrolysin vs 0.9% Saline Solution; The null-hypothesis stated no difference between the two treatment groups. A sample size of 103 evaluable patients per treatment group was estimated to allow for the detection of a significant group difference of 4.1 points in ADAS-cog+ weak 24 change score (standard deviation [SD] 9.0) in favor of Cerebrolysin with a power of 90% and a probability level of alpha-level 0.025 (one-sided); Test type: Superiority or Other; p < 0.0001, ANCOVA — P-value obtained from the F-test statistic of Cerebrolysin versus Placebo as part of ANCOVA (analysis of covariance). No adjustment for multiple comparisons was needed. The overall significance level alpha was fixed at alpha = 0.05 (two-sided); The study was designed to show significant differences in each of the two primary variables. No adjustment for multiple comparisons was needed; Mean Difference (Final Values) = -6.17, 95% CI 2-sided [-8.22 to -4.13]

2. Primary Outcome: CIBIC+ (Clinicians Interview-based Impression of Change) Score at Week 24
Description: This rating scale is based on the health care provider's "general clinical impressions" with the informant input (i.e. family members). It evaluates global function and is scored from 1 (marked improvement) to 7 (marked worsening).
Time Frame: week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Cerebrolysin | 0.9% Saline Solution
Number analyzed (Participants) | 117 | 115
Participants
  Marked improvement | 7 | 2
  Moderate improvement | 43 | 14
  Minimal improvement | 38 | 27
  No change | 20 | 52
  Minimal worsening | 9 | 16
  Moderate worsening | 0 | 4
  Marked worsening | 0 | 0

3. Secondary Outcome: Change From Baseline in ADAS-COG+ (Alzheimer's Disease Assessment Scale Cognitive Subpart)
Description: The modified Alzheimer's Disease Assessment Scale - Cognitive (ADAS-COG+) is a psychometric instrument used by a neuropsychologist that evaluates memory, attention, reasoning, language, orientation and praxis.
Time Frame: week 4, 12, 16
Reporting Status: Not Posted

4. Secondary Outcome: ADAS-COG+ Response
Description: A patient with an improvement from baseline of ≥ 4 points in the ADAS-COG+ score at a particular visit is considered to have an ADAS-COG+ response at that visit.
Time Frame: week 4, 12, 16, 24
Reporting Status: Not Posted

5. Secondary Outcome: Change From Baseline for Original ADAS-COG
Description: The Original Alzheimer's Disease Assessment Scale - Cognitive (ADAS-COG) is comprised of items 1-11 of the modified ADAS-COG+.
Time Frame: week 4, 12, 16, 24
Reporting Status: Not Posted

6. Secondary Outcome: CIBIC+ Score
Description: The Clinician Interview-based Impression of Change (CIBIC+) score is assigned by an experienced physician familiar with the manifestations of dementia after interviewing the patient and the caregiver.
Time Frame: week 4, 12, 16
Reporting Status: Not Posted

7. Secondary Outcome: CIBIC+ Response
Description: A patient with a CIBIC+ score of 1 to 3 at a particular visit is considered to have a CIBIC+ response at that visit. Patients with a score of 0, indicating that the assessment was not performed, are considered to be non-responders.
Time Frame: week 4, 12, 16, 24
Reporting Status: Not Posted

8. Secondary Outcome: CIBIS+ (Clinicians Interview-Based Impression of Severity)
Description: The Clinician Interview-based Impression of Disease Severity (CIBIS+) score is assigned by an experienced physician, familiar with the manifestations of dementia, after interviewing the patient and the caregiver.
Time Frame: week 24
Reporting Status: Not Posted

9. Secondary Outcome: Change From Baseline in MMSE (Mini-Mental State Examination) Score
Description: The Mini-Mental State Examination (MMSE) is a frequently used screening instrument for clinical trials conducted in patients with Alzheimer's Disease. It evaluates orientation, registration, attention and calculation, recall and language.
Time Frame: week 4, 12, 16, 24
Reporting Status: Not Posted

10. Secondary Outcome: Change From Baseline in ADCS-ADL (Alzheimer's Disease Cooperative Study-Activities of Daily Living Scale)
Description: The ADCS-ADL is a measure of functional disability. The ADCS-ADL assessment of activities of daily living is based on an interview with the caregiver.
Time Frame: week 4, 12, 16, 24
Reporting Status: Not Posted

11. Secondary Outcome: Change From Baseline in Trail-making Test
Description: The Trail-making test is a frequently used instrument for the assessment of executive function.
Time Frame: week 4, 12, 16, 24
Reporting Status: Not Posted

12. Secondary Outcome: Change From Baseline in Clock-drawing Test
Description: The Clock-drawing test is a frequently used screening instrument for dementia drug studies. It evaluates executive function of demented patients.
Time Frame: week 4, 12, 16, 24
Reporting Status: Not Posted

13. Secondary Outcome: Combined Response, i.e. Response in ADAS-COG+ and CIBIC+
Time Frame: week 4, 12, 16, 24
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Cerebrolysin | 0.9% Saline Solution
Serious Adverse Events (participants affected / at risk) | 3 | 0
Other Adverse Events (participants affected / at risk) | 0/117 | 0/115
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Cerebrolysin | 0.9% Saline Solution
Pyelonephritis acute (Infections and infestations) | 1/117 (1) | 0/115 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/117 (1) | 0/115 (0)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/117 (1) | 0/115 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No